CLINICAL TRIAL: NCT03575013
Title: A Phase 1b Study of Combination of Avelumab and Taxane Based Chemotherapy in Platinum Refractory or Ineligible Metastatic Urothelial Cancer
Brief Title: A Combination of Avelumab and Taxane (AVETAX) for Urothelial Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yousef Zakharia (Other)
Collaborators: Pfizer (Industry); University of Iowa (Other)
Responsible Party: Sponsor-Investigator, Yousef Zakharia, Clinical Associate Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201804833
Record Dates: First submitted 2018-06-18; First posted 2018-07-02 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-07

CONDITIONS: Urothelial Carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — avelumab; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Avelumab and Docetaxel (Experimental): Induction phase:
  Avelumab (10 mg/kg) + Docetaxel (75 mg/m2) every 3 weeks for 6 cycles
  Maintenance phase:
  Avelumab (10 mg/kg) every 2 weeks until disease progression or toxicity
  Interventions: Drug: Avelumab; Drug: Docetaxel

INTERVENTIONS:
Drug: Avelumab — Avelumab is a fully human anti-programmed death ligand 1 (PD-L1) IgG1 antibody
  Other Names: MSB0010718C
Drug: Docetaxel — Docetaxel is a antineoplastic agent belonging to the taxoid family
  Other Names: Taxotere

SUMMARY:
This study evaluates the safety and efficacy of the combination of Avelumab, (a fully human anti-programmed death ligand 1 (PD-L1) IgG1 antibody) in combination with a taxane chemotherapy (docetaxel) in patients with metastatic urothelial cancer who are either ineligible to receive cisplatin based chemotherapy, refractory to cisplatin in first line setting or have disease relapse after receiving cisplatin based chemotherapy within a year in the neoadjuvant or adjuvant setting.

DETAILED DESCRIPTION:
The study is a single institution, phase 1b, single arm non-randomized, open label prospective clinical trial to evaluate the combination of Avelumab and Docetaxel in adult subjects with locally advanced or metastatic urothelial carcinoma with disease progression during or following platinum-containing chemotherapy, or within 12 months of neoadjuvant or adjuvant platinum-containing chemotherapy.

The study has two phases:

1. A Phase 1b dose de-escalation of Docetaxel in combination with Avelumab, to establish the recommended phase 2 dose (RP2D) for the combination. The dose de-escalation phase will utilize a 3+3 design over 3 planned dose levels leading to the identification of a RP2D for the combination of Docetaxel and Avelumab. Note: Dose de-escalation is allowed only for Docetaxel and no changes will done to standard dose of Avelumab (i.e, 10 mg/kg).
2. In the dose expansion phase of the study, the fixed dose of Docetaxel in combination with Avelumab will be evaluated. The study is powered to a primary endpoint of overall response rate (ORR) with the combination of Docetaxel and Avelumab. Enrollment for part 2 will commence only after a RP2D is identified from phase 1.

ELIGIBILITY:
Inclusion Criteria:

* Age >/=18 years to 85 years
* Histologically or cytologically confirmed locally advanced or metastatic transitional cell carcinoma of the urothelium (including renal pelvis, ureters, urinary bladder, urethra). Additional mixed histologies such as squamous, plasmacytoid, adenocarcinoma, sarcomatoid, papillary, micropapillary are permitted provided the urothelial cancer is the predominant histological component.
* Eligible patients must have had either:

  * Progressed after treatment with at least 1 platinum-containing regimen, (e.g., ciplatin or carboplatin plus another agent such as gemcitabine, methotrexate, vinblastine, doxorubicin, etc.) for inoperable locally advanced or metastatic urothelial carcinoma or disease recurrence, or
  * Were ineligible for cisplatin-based chemotherapy, with ineligibility to cisplatin defined by impaired renal function (creatinine clearance < 60 ml/min), a hearing loss of 25 decibels at 2 contiguous frequencies, or grade ≥ 2 peripheral neuropathy or
  * Locally advanced or metastatic bladder cancer whose disease has progressed within 12 months of neoadjuvant or adjuvant chemotherapy.
* Biopsy material is required (archival tissue is acceptable if patient could not provide fresh or recent biopsy)
* ECOG performance status of 0 to 1
* Estimated life expectancy ≥3 months
* At least one measurable lesion by RECIST version 1.1
* Adequate hematologic function defined by white blood cell count ≥3 × 109/L with absolute neutrophil count ≥1.5 × 109/L, lymphocyte count ≥ 0.5 × 109/L, platelet count ≥100 × 109/L, and hemoglobin ≥9 g/dL (may have been transfused)
* Adequate hepatic function defined by a total bilirubin level ≤ the upper limit of normal range (ULN), an aspartate aminotransferase (AST) level ≤1.5 × ULN, and an alanine aminotransferase (ALT) level ≤1.5 × ULN
* Adequate renal function defined by an calculated creatinine clearance > 30 mL/min according to the Cockcroft-Gault formula
* Both male and female subjects must be willing to use highly effective contraception (that is, methods with a failure rate of less than 1% per year) throughout the study and for at least 30 days after last avelumab treatment administration if the risk of conception exists (see section 6.1.7). [NOTE: The effects of the study treatment on the developing human fetus are unknown; thus, women of childbearing potential and men must agree to use highly effective contraception, as stipulated in national or local guidelines. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, the treating physician should be informed immediately.
* Signed written informed consent

Exclusion Criteria:

* Concurrent treatment with an anticancer treatment
* Prior therapy with any drug targeting T cell coregulatory proteins
* Major surgery for any reason within 4 weeks or if the patient had not fully recovered within 4 weeks
* Concurrent systemic therapy with corticosteroids or other immunosuppressive agents, or use of any investigational drug within 28 days before starting trial drug; short-term administration of systemic steroids (that is, for allergic reactions or the management of immune-mediated adverse events while on study is allowed
* Patients with active central nervous metastases will be excluded. Appropriately treated CNS metastases with either surgery or radiation therapy are permitted to participate in the study
* Previous malignant disease (other than urothelial carcinoma) within the last 5 years, with the exclusion of basal or squamous cell carcinoma of the skin, cervical carcinoma in situ and prostate adenocarcinoma with Gleason score 6-7, pT2b.
* Prior organ transplantation, including allogenic stem-cell transplantation
* Known history of testing positive for HIV/AIDS, HBV, or HCV (including acute and chronic infection)
* Active or history of any autoimmune disease or immune-deficiencies (patients with type 1 diabetes, vitiligo, psoriasis, hypo- or hyperthyroid disease not requiring immunosuppressive treatment are eligible)
* Known monoclonal antibody hypersensitivity, history of anaphylaxis, or uncontrolled asthma
* Persisting toxicity related to prior therapy that was > grade 1 according to NCI-CTCAE v4.0; grade ≤2 sensory neuropathy is allowed
* Pregnancy or lactation
* Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure (≥ New York Heart Association Classification Class II), or serious cardiac arrhythmia requiring medication All other significant diseases, which in the investigator's opinion may influence the patient's tolerance of trial treatment. Other severe acute or chronic medical conditions including immune colitis, inflammatory bowel disease, immune pneumonitis, pulmonary fibrosis or psychiatric conditions including recent (within the past year) or active suicidal ideation or behavior; or laboratory abnormalities that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study
* Legal incapacity or limited legal capacity, including any psychiatric condition that would prohibit the understanding or rendering of informed consent
* Vaccination within 4 weeks of the first dose of Avelumab and while on study was prohibited except for administration of inactivated vaccines (e.g., inactivated influenza vaccines)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2018-10-29 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2024-02-09 (Actual)

PRIMARY OUTCOMES:
Dose De-Escalation Phase: To assess dose limiting toxicities (DLTs) using CTCAE v4.03. | From the start of treatment up to 5 years
  All adverse events (AEs )will be considered in DLT assessment unless an event is clearly unrelated to trial treatment. DLTs for phase 1b only include AEs that are considered possibly, probably, or definitely related to the Docetaxel plus Avelumab regimen which occur during the first 21 days of therapy. All AEs, including DLTs, are to be reported according to instructions in the Study Reference Manual and graded using the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03.
Dose Expansion Phase: To determine overall response rate (ORR) (complete response [CR] + partial response [PR]) per RECIST v1.1 | From the start of treatment up to 5 years
  Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 will be used to determine ORR.

SECONDARY OUTCOMES:
Dose Expansion: To determine radiologic progression-free survival (PFS) per RECIST v1.1 and immune RECIST criteria | From the start of treatment up to 5 years
  PFS is defined as the time between the first dose of study therapy and the earliest date of progression or death. Subjects who have neither progressed nor died will be censored at the last tumor assessment date for PFS.
Dose Expansion: To determine ORR per RECIST v1.1 | From the start of treatment up to 5 years
  Overall survival defined as the time between the first dose of study therapy and death (subjects who have not died will be censored at the most recent last-known-alive date).

CONTACTS AND LOCATIONS:
Overall Officials: Yousef Zakharia, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Garje R, Ravindra A, Rahim B, Kroll M, Johnson JS, Torres J, Bonner J, Packiam VT, Mott S, O'Donnell M, Zakharia Y. Avelumab and taxol chemotherapy in platinum-refractory or ineligible metastatic urothelial carcinoma (AVETAX trial). Urol Oncol. 2025 Sep;43(9):520.e9-520.e18. doi: 10.1016/j.urolonc.2025.04.005. Epub 2025 May 31. PMID 40451703

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-10-19): https://cdn.clinicaltrials.gov/large-docs/13/NCT03575013/Prot_SAP_000.pdf
  • Informed Consent Form (2021-01-12): https://cdn.clinicaltrials.gov/large-docs/13/NCT03575013/ICF_001.pdf